CLINICAL TRIAL: NCT03719222
Title: Analysis of Tumor Mutations and Tumor Microenvironment Using Archival Paraffin-embedded Tumor Specimens
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ACT Genomics (Industry)
Collaborators: Chi Mei Medical Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ACTG-18001
Record Dates: First submitted 2018-10-15; First posted 2018-10-25 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Sequence Analysis
Keywords: Genomic profiling assay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archived paraffin-embedded tumor specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non intervention — It is an non-interventional retrospective observational study by using archived paraffin-embedded tumor specimens

SUMMARY:
Genomic alterations have long been recognized as an important factor in tumor formation and drive tumor cell growth. However, the degree of genomic mutation (tumor mutation load, TMB) varies widely between tumors. In addition to gene mutations in tumor cells, the extent of immune cell infiltration in tumor tissues and the type and nature of immune cells (tumor microenvironment, TME) also play an important role in controlling tumor growth.

In recent years, more and more clinical studies have shown that the degree of genomic alteration (TMB) and tumor microenvironment (TME) have great potential in predicting a cancer patients' response to immunotherapy. Therefore, understanding the interaction and correlation between genomic alteration and tumor immune environment will not only deepen our understanding of tumor biology but also provide an important reference for developing immunotherapy treatment strategies for solid tumors.

DETAILED DESCRIPTION:
This is a non-interventional, mono-centric retrospective study to be carried out in Chi Mei Medical Center (CMMC) in order to determine the association between the genomic alterations and gene expression level of immune-related genes in cancer. Samples in paraffin-embedded block of biopsies or surgical pieces (either primary tumor or metastases) will be analyzed. For each sample, clinically relevant data associated with treated cancer and needed for characterization of tumor microenvironment will be documented. No additional procedures besides those already used in the routine clinical practice will be applied to the patients. Treatment assignment will be done according to the current practice.

This trial is, through accessing to archival tumor materials, to establish the relationship between tumor mutation burden and tumor immune microenvironment for future immunotherapy strategy.

ELIGIBILITY:
Inclusion Criteria:

* Sample from patients with histologically documented cancer in target population.

Exclusion Criteria:

* Unusable sample or biologically deteriorated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 600 cancer patients who fulfill the eligibiltiy criteria will be selected from the CMMC tissue bank. Eligible patients should have an available archival paraffin-embedded tumor block stored at the Department of Pathology, CMMC.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Correlation between TMB and the expression level of PD-1/PD-L1 | 12 months
  To explore possible relationship between genomic alteration and expression of immune-related genes in solid tumor, tumor mutation burden (TMB) and PD-1/PD-L1 expression level are examined and such relationship will be calculated by Pearson's correlation coefficient.

SECONDARY OUTCOMES:
Single point mutations, as part of cancer genomic profile | 12 months
  To establish a cancer genomic profile for the Asian population, genomic alterations such as point mutations will be assessed by NGS-based ACTOnco assay.
Small insertions and deletions (Indel), as part of cancer genomic profile | 12 months
  To establish a cancer genomic profile for the Asian population, genomic alterations such as small insertions and deletions will be assessed by NGS-based ACTOnco assay.
Copy number alterations, as part of cancer genomic profile | 12 months
  To establish a cancer genomic profile for the Asian population, genomic alterations such as copy number alterations will be assessed by NGS-based ACTOnco assay.
Microsatellite instability, as part of genomic profile | 12 months
  To establish a cancer genomic profile for the Asian population, genomic alterations such as microsatellite instability will be assessed by NGS-based ACTOnco assay.
TME gene expression profile, which consists of quantitative measurements of immune-related genes | 12 months
  To establish an expression signature of tumor microenvironment (TME) in addition to PD-1 and PD-L1, >90 immune-related genes will be assessed by ACTTME assay via quantitative PCR
Concordance of TMB between ACTOnco assay and an externally validated assay | 12 months
  To compare between calculated tumor mutation burden values (TMB, in mutations per megabase) resulting from different methodologies, concordance between two NGS-based assays will be expressed as positive predictive value (PPV) and negative predictive value (NPV).

CONTACTS AND LOCATIONS:
Locations (1):
- ACT Genomics, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No